CLINICAL TRIAL: NCT03477721
Title: The Role of the Muscle-nervous System Interface in Cancer Cachexia
Acronym: NUMANCAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Laviano, Alessandro Laviano, MD associate professor of Internal Medicine, University of Roma La Sapienza
Other Study IDs: NUMANCAN
Record Dates: First submitted 2018-03-11; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cachexia; Cancer; Sarcopenia
Keywords: Agrin Fragment C-terminus (CAF)
MeSH Terms: conditions — Cachexia; Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples: determination of: serum C-reactive protein, albumin, creatinine and haemoglobin concentrations. Agrin fragment c-terminus and IL-6 will be carried out using specific ELISA kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with cancer cachexia (CTB): For diagnosis of cachexia it will be used the following criteria (Evans et al., 2008)
- Group without cancer cachexia (TB)

SUMMARY:
Sarcopenia is an important component of cachexia associated with cancer, and their high incidence in cancer patients emphasizes the need for a better understanding of its mechanisms, which can result in better therapeutic interventions to reverse this situation and improve the prognosis. Our hypothesis is that the plasma concentration of IL-6 and c-terminal agrin is directly correlated with the loss of muscle mass and development of cachexia.

DETAILED DESCRIPTION:
The agrin is a protein that acts on neuromuscular junctions (NMJs) promoting stabilization of same, which results in the maintenance and growth of muscle fibers, but the cleavage of agrin, a process by which is formed the agrin fragment C-terminus (CAF), has been linked to the development of sarcopenia, because its presence is directly linked to the reduction in the number of muscle fibers, increasing the heterogeneity of fiber size, presence of Central cores and increasing the proportion of type I fibers and consequently a greater degradation of lean body mass. Studies in mice show that the greatest cleavage of agrin carries on development of sarcopenia and human studies report that individuals with higher serum levels of sarcopenia CAF compared to individuals without sarcopenia.

Therefore, aiming at the complexity of cancer associated with the cachexia and the great importance of the maintenance of lean body mass to a better prognosis in disease, is of fundamental importance to elucidate the role of CAF and the factors associated with sarcopenia, the possible use of these proteins for diagnosis and the contribution that this clarification could bring in clinical therapy.

ELIGIBILITY:
Inclusion Criteria:

* cancer diagnosis

Exclusion Criteria:

* continuously use of anti-inflammatory medications;
* present renal and/or liver failure,
* AIDS,
* inflammatory bowel disease or chronic inflammatory processes not related to cachexia.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Oure sample will be selected between cancer patient of Rome Umberto I Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-04-16 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Agrin fragment c-terminus CAF in cancer and cancer cachexia | 1 month
  To measure the contents of agrin fragment c-terminus (CAF) in plasma of patient with cancer and cancer cachexia.
Agrin fragment c-terminus CAF in cancer sarcopenia | 1 month
  To analyze correlation between Agrin fragment c-terminus CAF and the lean body mass (CT-scan estimated) of patients with cancer and with cancer cachexia.
Agrin fragment c-terminus CAF and IL-6 levels | 1 month
  To correlate levels of agrin fragment c-terminus (CAF) and IL-6 plasma levels in patients with cancer and with cancer cachexia.
Agrin fragment c-terminus (CAF) and IL-6 and lean body mass | 1 month
  To correlate levels of agrin fragment c-terminus (CAF) and IL-6 with the lean body mass

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Laviano, MD, Principal Investigator — Department of Clinical Medicine, Sapienza University of Rome, Italy
Locations (1):
- Department of Clinical Medicine, Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We are still evaluate a researcher to analyze data collected

REFERENCES:
- [Background] Argiles JM, Alvarez B, Lopez-Soriano FJ. The metabolic basis of cancer cachexia. Med Res Rev. 1997 Sep;17(5):477-98. doi: 10.1002/(sici)1098-1128(199709)17:53.0.co;2-r. No abstract available. PMID 9276862
- [Background] Argiles JM, Busquets S, Toledo M, Lopez-Soriano FJ. The role of cytokines in cancer cachexia. Curr Opin Support Palliat Care. 2009 Dec;3(4):263-8. doi: 10.1097/SPC.0b013e3283311d09. PMID 19713854
- [Background] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Background] Batista ML Jr, Peres SB, McDonald ME, Alcantara PS, Olivan M, Otoch JP, Farmer SR, Seelaender M. Adipose tissue inflammation and cancer cachexia: possible role of nuclear transcription factors. Cytokine. 2012 Jan;57(1):9-16. doi: 10.1016/j.cyto.2011.10.008. Epub 2011 Nov 17. PMID 22099872
- [Background] Belizario JE, Fontes-Oliveira CC, Borges JP, Kashiabara JA, Vannier E. Skeletal muscle wasting and renewal: a pivotal role of myokine IL-6. Springerplus. 2016 May 13;5:619. doi: 10.1186/s40064-016-2197-2. eCollection 2016. PMID 27330885
- [Background] Evans WJ, Morley JE, Argiles J, Bales C, Baracos V, Guttridge D, Jatoi A, Kalantar-Zadeh K, Lochs H, Mantovani G, Marks D, Mitch WE, Muscaritoli M, Najand A, Ponikowski P, Rossi Fanelli F, Schambelan M, Schols A, Schuster M, Thomas D, Wolfe R, Anker SD. Cachexia: a new definition. Clin Nutr. 2008 Dec;27(6):793-9. doi: 10.1016/j.clnu.2008.06.013. Epub 2008 Aug 21. PMID 18718696
- [Background] Fan Y, Mao R, Yang J. NF-kappaB and STAT3 signaling pathways collaboratively link inflammation to cancer. Protein Cell. 2013 Mar;4(3):176-85. doi: 10.1007/s13238-013-2084-3. Epub 2013 Mar 13. PMID 23483479
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Fearon KC, Moses AG. Cancer cachexia. Int J Cardiol. 2002 Sep;85(1):73-81. doi: 10.1016/s0167-5273(02)00235-8. PMID 12163211
- [Background] Fearon KC, Voss AC, Hustead DS; Cancer Cachexia Study Group. Definition of cancer cachexia: effect of weight loss, reduced food intake, and systemic inflammation on functional status and prognosis. Am J Clin Nutr. 2006 Jun;83(6):1345-50. doi: 10.1093/ajcn/83.6.1345. PMID 16762946
- [Background] Gonzalez-Freire M, de Cabo R, Studenski SA, Ferrucci L. The Neuromuscular Junction: Aging at the Crossroad between Nerves and Muscle. Front Aging Neurosci. 2014 Aug 11;6:208. doi: 10.3389/fnagi.2014.00208. eCollection 2014. PMID 25157231
- [Background] Hettwer S, Dahinden P, Kucsera S, Farina C, Ahmed S, Fariello R, Drey M, Sieber CC, Vrijbloed JW. Elevated levels of a C-terminal agrin fragment identifies a new subset of sarcopenia patients. Exp Gerontol. 2013 Jan;48(1):69-75. doi: 10.1016/j.exger.2012.03.002. Epub 2012 Mar 11. PMID 22433628
- [Background] Kalinkovich A, Livshits G. Sarcopenia--The search for emerging biomarkers. Ageing Res Rev. 2015 Jul;22:58-71. doi: 10.1016/j.arr.2015.05.001. Epub 2015 May 8. PMID 25962896
- [Background] Kern KA, Norton JA. Cancer cachexia. JPEN J Parenter Enteral Nutr. 1988 May-Jun;12(3):286-98. doi: 10.1177/0148607188012003286. PMID 3292798
- [Background] Kujawski M, Kortylewski M, Lee H, Herrmann A, Kay H, Yu H. Stat3 mediates myeloid cell-dependent tumor angiogenesis in mice. J Clin Invest. 2008 Oct;118(10):3367-77. doi: 10.1172/JCI35213. PMID 18776941
- [Background] Kumar NB, Kazi A, Smith T, Crocker T, Yu D, Reich RR, Reddy K, Hastings S, Exterman M, Balducci L, Dalton K, Bepler G. Cancer cachexia: traditional therapies and novel molecular mechanism-based approaches to treatment. Curr Treat Options Oncol. 2010 Dec;11(3-4):107-17. doi: 10.1007/s11864-010-0127-z. PMID 21128029
- [Background] Mantovani A, Allavena P, Sica A, Balkwill F. Cancer-related inflammation. Nature. 2008 Jul 24;454(7203):436-44. doi: 10.1038/nature07205. PMID 18650914
- [Background] Mignogna MD, Fedele S, Lo Russo L, Lo Muzio L, Bucci E. Immune activation and chronic inflammation as the cause of malignancy in oral lichen planus: is there any evidence ? Oral Oncol. 2004 Feb;40(2):120-30. doi: 10.1016/j.oraloncology.2003.08.001. PMID 14693234
- [Background] Okada F. Inflammation-related carcinogenesis: current findings in epidemiological trends, causes and mechanisms. Yonago Acta Med. 2014 Jun;57(2):65-72. Epub 2014 Jul 30. PMID 25324587
- [Background] Roxburgh CS, McMillan DC. Cancer and systemic inflammation: treat the tumour and treat the host. Br J Cancer. 2014 Mar 18;110(6):1409-12. doi: 10.1038/bjc.2014.90. Epub 2014 Feb 18. PMID 24548867
- [Background] Scherbakov N, Knops M, Ebner N, Valentova M, Sandek A, Grittner U, Dahinden P, Hettwer S, Schefold JC, von Haehling S, Anker SD, Joebges M, Doehner W. Evaluation of C-terminal Agrin Fragment as a marker of muscle wasting in patients after acute stroke during early rehabilitation. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):60-7. doi: 10.1002/jcsm.12068. Epub 2015 Oct 27. PMID 27066319
- [Background] Tisdale MJ. Cancer cachexia. Curr Opin Gastroenterol. 2010 Mar;26(2):146-51. doi: 10.1097/MOG.0b013e3283347e77. PMID 19918173
- [Background] Srdic D, Plestina S, Sverko-Peternac A, Nikolac N, Simundic AM, Samarzija M. Cancer cachexia, sarcopenia and biochemical markers in patients with advanced non-small cell lung cancer-chemotherapy toxicity and prognostic value. Support Care Cancer. 2016 Nov;24(11):4495-502. doi: 10.1007/s00520-016-3287-y. Epub 2016 May 28. PMID 27236439